CLINICAL TRIAL: NCT04884139
Title: DTG/3TC vs. BIC/FTC/TAF Maintenance Therapy in People Living With HIV: an Open-label Randomized Clinical Trial
Brief Title: DTG/3TC vs. BIC/FTC/TAF Maintenance Therapy in People Living With HIV:
Acronym: PASO-DOBLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA11720
Record Dates: First submitted 2021-05-05; First posted 2021-05-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — dolutegravir; Lamivudine; bictegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dovato arm (Experimental): DTG/3TC
  Interventions: Drug: Dolutegravir/Lamivudine as a single pill
- Biktarvy arm (Active Comparator): BIC/FTC/TAF
  Interventions: Drug: Bictegravir/Emtricitabine/Tenofovir alfenamide as a single pill.

INTERVENTIONS:
Drug: Dolutegravir/Lamivudine as a single pill — - Dose: Dolutegravir 50mg/ Lamivudine 300 mg -Route of adminstration: oral -Schedule of administration: once a day for 96 weeks.
  Arms: Dovato arm
Drug: Bictegravir/Emtricitabine/Tenofovir alfenamide as a single pill. — * Dose: Bictegravir 50 mg/Emtricitabine 200 mg /Tenofovir alafenamide 25 mg
  * Route of adminstration: oral
  * Schedule of administration: once a day for 96 weeks.
  Arms: Biktarvy arm

SUMMARY:
The hypothesize that DTG/3TC will be non-inferior to BIC/FTC/TAF with a 4% margin in virologically suppressed HIV-infected patients. The study will allow claiming for Superiority. Assuming that both DTG and BIC may lead to similar weight gains (approximately 1 kg after 48 weeks) in virologically suppressed HIV-infected patients and that TAF may induce a further weight gain (approximately 1 kg after 48 weeks), also hypothesize that switching to BIC/FTC/TAF may lead to greater weight gain than switching to DTG/3TC over 48 weeks.

This trial is a Phase IV, open-label, randomized multicentre clinical trial evaluating the efficacy of DTG/3TC versus BIC/FTC/TAF for the maintenance of virological suppression in HIV patients.

DETAILED DESCRIPTION:
Participants will be randomly assigned in a 1:1 ratio to receive DTG/3TC or BIC/FTC/TAF. Randomization will be stratified by sex and TAF use at baseline. At least 33% of the patients included will be women.

The investigator will also endeavour to recruit as many non-Caucasian participants as possible.

Patients with TAF-containing regimens at baseline will be limited to 25% or less of the total number of participants.

Three sub-studies will be performed: Omics sub-study ; Senescence sub-study; Fat biopsies sub-study.

Omics sub-study: Assess the mechanistic pathways involved on weight changes associated with switching to BIC/FTC/TAF vs. DTG/3TC.

Senescence sub-study: Assess the potential effects on the telomere length, epigenetic age and oxidative stress markers of switching to BIC/FTC/TAF vs. DTG/3TC.

Fat biopsies sub-study: To assess potential effects of switching to BIC/FTC/TAF vs.

DTG/3TC on expression of marker genes of mitochondrial function, adipogenesis, and inflammation in subcutaneous fat tissue. Assays on adipose tissue gene expression will be complemented by analysis in serum of adipokines representative of adipose tissue function (leptin, adiponectin), and inflammation biomarkers (TNFalpha, MCP-1, IL-6, IL-8, IL-10, IL-18).

ELIGIBILITY:
Inclusion Criteria:

1. Understanding the study information provided and being capable of giving written informed consent.
2. Confirmed HIV infection.
3. ≥18 years of age on the day of screening.
4. HIV RNA <50 copies/mL for at least 24 weeks before screening.
5. Receiving any regimen for HIV containing more than 1 pill a day or any single tablet regimen containing at least one of the following: cobicistat-boosting, efavirenz, or tenofovir disoproxyl fumarate, for at least 24 weeks before screeningPatients with TAF are expected from cobiscitat-boosting single tablet regimens containing darunavir or elvitegravir and from more-than-1-pill-a-day regimens containing TAF/FTC; their participation will be limited to ≤25%. Patients will be stratified according to the presence or not of TAF in their regimens.
6. No evidence of previous viral failure.
7. No known or suspected resistance to study drugs.
8. Females of childbearing potential, must be using highly effective methods of contraception from study inclusion and for at least 4 weeks after last study visit; all female volunteers must be willing to undergo urine pregnancy testing at the time points specified in the schedules of events.
9. Clinical stability: Participants who are healthy (other than HIV infection) as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, laboratory tests, and cardiac monitoring.

Exclusion Criteria:

1. Is pregnant or lactating at the screening visit or at any time during the study or is planning on becoming pregnant over the duration of the study.
2. Evidence of Hepatitis B virus infection based on at least one positive result of testing at Screening for Hepatitis B surface antigen (HBsAg) and Hepatitis B core antibody (anti- HBc).
3. Previous or current therapy with dolutegravir or bictegravir.
4. History of allergy to study drugs or their components.
5. Liver disease as defined by ALT >= 5x ULN or ALT >=3xULN and Bili =1.5xULN (with >35% direct bilirubin).
6. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (apart from hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones);
7. Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification and/or anticipated need for Hep C treatment.
8. Kidney disease as defined by CKD-EPI <50ml/min.
9. Any recently (<=6 months) diagnosed clinical condition or recently (<=6 months) initiated concomitant therapy (see Section 6.5) that may primarily affect weight or body composition. E.g., including but not limited to endocrine disorders, osteoporosis or medications to treat these clinical conditions, with the exception of ontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA ≥50 copies/mL | Week 48

SECONDARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA ≥50 copies/mL | week 96
Proportion of patients with plasma HIV-1 RNA <50 copies/mL | Week 48 and week 96
Absolute weight | Basal, week 48 y week 96
BMI change | Basal, week 48 y week 96
Proportion of patients with weight change >5% | Basal, week 48 y week 96
Absolute values in CD4+ cells count | Basal, week 48 y week 96
Changes in CD4+ cells count | Basal, week 48 y week 96
Absolute values CD4:CD8 ratio | Basal, week 48 y week 96
Changes CD4:CD8 ratio | Basal, week 48 y week 96
Change in total and regional (trunk and extremities) fat by DXA | Basal, week 48 y week 96
Change in total and regional (trunk and extremities) fat-free mass by DXA | Basal, week 48 y week 96
Change in lumbar and hip bone mineral density (BMD) by DXA | Basal, week 48 y week 96
Change trabecular bone score (TBS) by DXA | Basal, week 48 y week 96
Change in subcutaneous and visceral fat (CT) | Basal, week 48 y week 96
Change in fasting glucose cholesterol, triglycerides), and FIB-4 score | Basal, week 48 y week 96
Change insulin cholesterol, triglycerides), and FIB-4 score | Basal, week 48 y week 96
Change in HOMA-IR cholesterol, triglycerides), and FIB-4 score | Basal, week 48 y week 96
Change in HbA1c cholesterol, triglycerides), and FIB-4 score | Basal, week 48 y week 96
Change in plasma lipids (total, HDL, and LDL) cholesterol, triglycerides), and FIB-4 score | Basal, week 48 y week 96
Changes in estimated glomerular filtration rate (CKD-EPI) | Basal, week 48 y week 96
Changes in urinary protein/creatinine | Basal, week 48 y week 96
Change in blood pressure | Basal, week 48 y week 96
  Systolic and Diastolic Blood Pressure
Change in sleep quality (Pittsburg Sleep Quality Index) | From basal, until week 96 , in each visit
  Pittsburg Sleep Quality Index
Change in anxiety and depression (HAD) quality of life (HIV Symptom Index questionnaire / Symptom Distress Module (HIV-SI/SDM | From basal, until week 96 , in each visit
  Anxiety and depression (HAD) questionnaire
Change in quality of life (HIV Symptom Index questionnaire / Symptom Distress Module (HIV-SI/SDM) | From basal, until week 96 , in each visit
  Quality of life (HIV-SI/SDM) questionnaire
Incidence and severity of adverse events (clinical and laboratory) | From basal, until week 96 , in each visit
Incidence of adverse events leading to treatment discontinuation. | From basal, until week 96 , in each visit
Incidence of genotypic resistance mutations in participants with virological failure | Week 48 and week 96

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Martinez, MD, Principal Investigator — H. Clinc de Barcelona
Locations (33):
- Spain (33):
  - H. Marina Baixa, Villajoyosa, Alicante
  - Hospital Fundación Alcorcón, Alcorcón, Madrid
  - CHUAC, A Coruña
  - H. General Universitario Dr. Balmis, Alicante
  - H. de Elche, Alicante
  - H. de Torrecárdenas, Almería
  - H. Clinic, Barcelona
  - H. Germans Trias i Pujol, Barcelona
  - H. de Bellvitge, Barcelona
  - H. de Igualada, Barcelona
  - H. del Mar, Barcelona
  - H. San Joan de Deu, Barcelona
  - H. Sant Creu y Sant Pau, Barcelona
  - H. Vall de Hebron, Barcelona
  - H. Universitario de Guadalajara, Guadalajara
  - H. Juan Ramón Jimenez, Huelva
  - Hospital Universitari Arnau de Vilanova, Lleida
  - H. Infanta Leonor, Madrid
  - H. La Princesa, Madrid
  - H. Príncipe de Asturias, Madrid
  - H. Univ. La Paz, Madrid
  - H. Univ. Puerta de Hierro, Madrid
  - H. Costa del Sol, Marbella
  - H. Reina Sofía, Murcia
  - H. Central de Asturias, Oviedo
  - H. Son Espases, Palma de Mallorca
  - H. Son Llatzer, Palma de Mallorca
  - H. de Valme, Seville
  - H. Joan XXIII, Tarragona
  - H. Clínico Univ. de Valencia, Valencia
  - H Clinico Univ. de Valladolid, Valladolid
  - H. Alvaro Cunquerio, Vigo
  - H. Clinico Univ. Lozano Bleza, Zaragoza

REFERENCES:
- [Derived] Ryan P, Blanco JL, Masia M, Garcia-Fraile L, Crusells MJ, Domingo P, Curran A, Guerri-Fernandez R, Bernal E, Bravo J, Revollo B, Macias J, Tiraboschi JM, Montejano R, Amador C, Torralba M, Merino D, Diaz-Brito V, Galindo MJ, Ferra S, Villoslada A, Losa JE, Fanjul FJ, Perez-Stachowski X, Peraire J, Portilla J, de la Fuente S, Duenas C, Vazquez MJ, Di Gregorio S, Esteban H, Gil P, de Miguel M, Alejos B, Martinez E; PASO-DOBLE study group. Maintenance therapy with dolutegravir and lamivudine versus bictegravir, emtricitabine, and tenofovir alafenamide in people with HIV (PASO-DOBLE): 48-week results from a randomised, multicentre, open-label, non-inferiority trial. Lancet HIV. 2025 Jul;12(7):e473-e484. doi: 10.1016/S2352-3018(25)00105-5. Epub 2025 Jun 7. PMID 40489982